CLINICAL TRIAL: NCT06625229
Title: Fourth Generation Percutaneous Transverse Osteotomies for Hallux Valgus
Status: Completed | Type: Observational
Sponsor: Orthopaedic and Arthritis Specialist Centre (Other)
Responsible Party: Principal Investigator, Thomas Lewis, Principal Investigator, Orthopaedic and Arthritis Specialist Centre
Other Study IDs: PLHV2024
Record Dates: First submitted 2024-09-20; First posted 2024-10-03 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-10

CONDITIONS: Hallux Valgus Deformity; Hallux Valgus (Bunion) Resection; Hallux Valgus Surgery; Hallux Deformity; Forefoot Surgery; Minimally Invasive Surgical Procedures; Minimally Invasive Surgical Technique; Hallux Abductovalgus
Keywords: Bunion; Hallux valgus; percutaneous surgery; minimally invasive surgery; forefoot deformity; metatarsal osteotomy; patient reported outcome measure; Manchester Oxford Foot Questionnaire (MOXFQ); Osteotomy; Observational Study
MeSH Terms: conditions — Hallux Valgus; Bunion

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Consecutive patients: Consecutive patients aged 16 years and over, who had exhausted conservative treatment and subsequently underwent primary correction of hallux valgus (of any deformity severity) were included. Patients who underwent additional forefoot procedures eg. hammer toe corrections, distal metaphyseal metatarsal osteotomy, were included. Patients who had previously had hallux valgus surgery, or first ray degenerative joint disease were excluded.

SUMMARY:
The goal of this observational study is to learn if percutaneous transverse osteotomies for hallux valgus deformity are safe and effective. The main questions it aims to answer are:

1. What is the change in clinical patient reported outcome measures after minimally invasive bunion surgery
2. What severity of bunion deformity can be corrected with minimally invasive surgery
3. What factors may lead to recurrence of bunion deformity
4. What is the rate of complications following bunion deformity surgery

Researchers will retrospectively review a research registry containing prospectively collected clinical and radiographic deformity data collected as part of routine care.

ELIGIBILITY:
Inclusion Criteria:

* Primary diagnosis of hallux valgus that has failed conservative treatment

Exclusion Criteria:

* Degenerative changes of first MTPJ
* Previous hallux valgus deformity correction surgery

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Consecutive patients presenting to a private surgeon in Sydney, Australia
Sampling Method: Non-Probability Sample
Enrollment: 483 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Manchester-Oxford Foot Questionnaire (MOXFQ) | Patients completed the MOXFQ at 6,12 and 24 months following surgery. Patients outside of these time points were asked to complete scores at their final follow up.
  A validated patient reported outcome measure for assessment of function in hallux valgus.
  The Manchester Oxford Foot Questionnaire (MOXFQ) consists of 3 domains (walking and standing, social interaction [based on the patient's self-consciousness regarding their feet/shoes as well as the overall impact on social, recreational, work, and other everyday activities], and pain), with the score in each domain ranging from 0 (best possible score) to 100 (worst possible score). An overall summary "index" score can also be calculated. The minimal clinically important difference (MCID) has been shown to be 16, 12, and 24 for the walking and standing, pain, and social interaction domains, respectively.

SECONDARY OUTCOMES:
Complication Data | Clinical notes were reviewed at final follow up (minimum 12 months post surgery) following surgery to assess for any complications
  Complication data were routinely prospective collected for all patients until discharge and categorised using a modified Clavien-Dindo complication classification.
EuroQol 5D Health Related Quality of Life (EQ-5D) | Patients completed the EQ5D at 6,12 and 24 months following surgery. Patients outside of these time points were asked to complete scores at their final follow up(minimum 12 months following surgery).
  A validated patient reported outcome measure for health related quality of life. The EQ-5D is a standardized patient-reported outcome measure (PROM) assessing health across five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has five levels of severity, from no problems to extreme problems. The scores are combined into a health profile and converted into a single index value reflecting overall health, where 1 represents perfect health, 0 represents death, and negative values indicate health states worse than death. The EQ-5D also includes a visual analog scale (VAS) for patients to rate their overall health.
Radiographic Deformity Correction | Specified timepoints during study (6weeks, 6months, final follow up (minimum 12 months following surgery)
  The intermetatarsal angle (IMA) and hallux valgus angle (HVA) were measured according to the American Orthopaedic Foot &amp; Ankle Society technique and categorised with regards to deformity severity. pre-operatively, six months following surgery and final follow up. Round sign and sesamoid coverage were classified according to Okuda et al. and Yildirim et al.
Visual Analogue Scale for Pain (VAS Pain) | Patients completed the VAS Pain at 6,12 and 24 months following surgery. Patients outside of these time points were asked to complete scores at their final follow up(minimum 12 months following surgery).
  A validated outcome measure to assess pain. The Visual Analog Scale (VAS) for pain consists of a straight line with one end labeled no pain(0) and the other worst possible pain(100). Patients mark a point on the line that represents their pain level, and the distance from the no pain end to the mark is measured to quantify the pain. Higher scores indicate greater pain intensity, with 0 being no pain and 100 being the worst imaginable pain.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Lam, MBBS (Hons), FRACS,, Principal Investigator — Orthopaedic and Arthritis Specialist Centre, Chatswood, Sydney, Australia
Locations (1):
- Orthopaedic and Arthritis Specialist Centre, Sydney, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: No
Patient consent not discussed for sharing of IPD